CLINICAL TRIAL: NCT05180643
Title: Exploratory Feasibility Study for the Development of Mindfulness-based Stress Reduction Program (MBSR )in Parkinsonian Patients - MPARK
Brief Title: Mindfulness Meditation (MBSR) and Parkinson's Disease (PD)
Acronym: M-PARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2019/32
Record Dates: First submitted 2020-02-06; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson; MBSR; Mindfulness
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This is a prospective exploratory monocentric pilot study in the context of interventional research with minimal risks and constraints, which aims to collect qualitative and quantitative data from two pilot 8-week MBSR programs organized at the University Hospital Center. Bordeaux with two groups of patients: 10 non-fluctuating patients or with minor fluctuations (Group A) and 10 patients with mild to moderate fluctuations (Group B).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-fluctuating patients or with minor fluctuations (Group A) (Experimental): Patient without fluctuation or with minor motor fluctuations (rated 0 or 1 on all 5 items of the UPDRS-dyskinesia and Motor Fluctuations scale)
  Interventions: Behavioral: Mindfulness-Based Stress Reduction-based program (MBSR).
- patients with mild to moderate fluctuations (Group B). (Experimental): Patient without fluctuation or with minor to moderate motor fluctuations (rated 2 or 3 on all 5 items of the UPDRS-dyskinesia and Motor Fluctuations scale)
  Interventions: Behavioral: Mindfulness-Based Stress Reduction-based program (MBSR).

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction-based program (MBSR). — The MBSR program is built over 8 weeks (1 information session, 8 group sessions from 2h30 to 3h and 1 full day). A trained MBSR instructor will lead group sessions weekly for approximately 150-210 minutes to teach and demonstrate the practices. Practices include walking/standing/supine meditation, body scanning (drawing attention to various areas of the body such as the right foot or left hand), and simple hatha yoga postures. Exercises are the basis of this group learning with practice time and practice exchange time. Participants are asked to commit to daily meditation at home using audioguides for 40 minutes to 1 hour.

SUMMARY:
Non-pharmacological therapies become more important in the management of Parkinson's disease (PD). Among these, mindfulness meditation is the subject of high expectations. This intervention, such as the Mindfulness-Based Stress Reduction-based (MBSR) stress reduction program, have shown effects on psychological distress, motor and non-motor disorders, and quality of life. However, the data is still very frail and the conditions for practical use are still very uncertain. The objective of the study is to determine the feasibility of a standardized MBSR program in Parkinsonians patients.

DETAILED DESCRIPTION:
Recent interest has developed in non-drug methods in the management of PD, especially for non-motor signs since recent years. Numerous studies have been investigated this issue, particularly in regard to mindfulness meditation approaches. Nowadays, the mindfulness-based stress reduction program (MBSR) is the most studied in medicine ([18]). The MBSR program has been studied in Parkinson's disease in numerous studies ([24], [3], [1], [9]) and the program compliance is reported as variable,from high (80%, [24], [9]) to modest (50%,; [3]), with little data on acceptability. Mindfulness meditation in the management of Parkinson's disease is the subject of high expectations for patients and their caregivers but the scientific literature is still very frail and the conditions for practical use in our country remains still very uncertain. What is the feasibility and acceptability of a standard MBSR-type program? For which type of patients? For which symptom (s)? What are the benefits, constraints and / or adverse effects felt? If a nationwide interventional trial were to be proposed, what would be the primary objective? What would be the ideal design? The MBSR program is a standardized group program (10 to 20 people) over 8 weeks. The program is progressive and structured, essentially practical, participatory and interactive, encouraging and supportive. The MBSR program will be supplemented by two visits (1 month before and 1 month later) including: a global clinical evaluation (MDS-UPDRS), a cognitive evaluation (MOCA and TAP battery), depression (BDI-II) and anxiety scales (PAS, self-questionnaire), sleep (Pittsburgh Sleep Quality Index), pain (EVA) and quality of life (PDQ-39). In addition, a qualitative interview on the expectations of the program will be carried during the pre-program interview and a qualitative descriptive evaluation on the acceptability, the adverse effects and the feeling of the program during the post-program interview.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with Parkinson's disease
* Aged over 18
* Under 80 years old
* Patient without fluctuation or with minor to moderate motor fluctuations (rated 0 or 3 on all 5 items of the UPDRS-dyskinesia and Motor Fluctuations scale)
* Patient with Hoehn Stadium and Yahr from 1 to 3
* Patient not presenting with acute depression not stabilized by the treatment or during the last 6 months
* Patient without unstable psycho-behavioral disorders (hallucinations, psychoses, impulse control disorders) less than 6 months
* Patient affiliated or beneficiary of the social security scheme
* Free, informed and written consent (at the latest on the day of inclusion and before any research required by the research).

Exclusion Criteria:

* Patient with Hoehn Stadium and Yahr over 3
* Patient with major cognitive impairment (MOCA <24)
* Patient with severe motor fluctuation (rated> 3 for all 5 items on the dyskinesia MDS-UPDRS scale and Motor Fluctuations)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
the rate of patients who completed the entire MBSR program | 6 months after inclusion
  the rate of patients who completed the meditation sessions, the full meditation day, and one-to-one daily compliance rate

SECONDARY OUTCOMES:
Achievement of the MBSR (Mindfulness Based Stress Reduction) program from individual pre-program interview | the pre-program interview will be performed 2 months after inclusion (one month before the MBSR program's beginning)
  Failure factors, problems encountered determined from a individual pre-program interview lasting about 20 minutes for achievement of the MBSR program request
Achievement of the MBSR (Mindfulness Based Stress Reduction) program from individual post-program interview | the post-program interview will be performed 6 months after inclusion (one month after the end MBSR program)
  Failure factors, problems encountered determined from a individual post-program interview lasting about 20 minutes for achievement of the MBSR program request
Acceptability of the MBSR (Mindfulness Based Stress Reduction) program from individual pre-program interview | the pre-program interview will be performed 2 months after inclusion ( one month before the MBSR program's beginning) and will last about one hour in total
  Program compliance for collective and individual meditations determined from a individual pre-program interview lasting about 20 minutes for acceptability of the MBSR program request
Acceptability of the MBSR (Mindfulness Based Stress Reduction) program from individual post-program interview | the post-program interview will be performed 6 months after inclusion (one month after the end MBSR program)
  Program compliance for collective and individual meditations determined from a individual post-program interview lasting about 20 minutes for acceptability of the MBSR program request
Expectations with regard to the MBSR (Mindfulness Based Stress Reduction) program determined from individual pre-program interview | the pre-program interview will be performed 2 months after inclusion ( one month before the MBSR program's beginning)
  Patient feelings, impressions and attitudes towards the program determined from a individual pre-program interview lasting about 20 minutes for expectations with regard to the MBSR program request
Expectations with regard to the MBSR (Mindfulness Based Stress Reduction)program determined from individual post-program interview | the post-program interview will be performed 6 months after inclusion ( one month after the MBSR program's beginning)
  Patient feelings, impressions and attitudes towards the program determined from a individual post-program interview lasting about 20 minutes for the request on expectations with regard to the MBSR program
Motor and non-motor symptoms evaluated by the MDS-UPDRS (Unified Parkison's Disease Ratinf Scale) score at the inclusion | at enrollment
  The MDS-UPDRS score is based on the "Unified Parkinson's Disease Rating Scale" : the MDS-UPDRS makes it possible to assess the different motor and non-motor symptoms. The MDS-UPDRS has four parts: Non-motor experiences of daily life (13 questions); Motor experiences of daily life (13 questions); Motor exam (18 items); Motor complications (6 items). All items are scored from 0 to 4 and are clearly defined: 0: normal, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe. The duration of the exam is 10 minutes.
Motor and non-motor symptoms evaluated by the MDS-UPDRS (Unified Parkison's Disease Ratinf Scale) score at the end of the following period | at the end of the following period ( i.e. 6 months after the inclusion, 1 month after the end of the MBSR program
  The MDS-UPDRS score is based on the "Unified Parkinson's Disease Rating Scale": The MDS-UPDRS has four parts: Non-motor experiences of daily life (13 questions); Motor experiences of daily life (13 questions); Motor exam (18 items); Motor complications (6 items). All items are scored from 0 to 4 and are clearly defined: 0: normal, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe. The duration of the exam is 10 minutes.
Cognitive efficiency evaluated by the "Montreal Cognitive Assessment" (MOCA) at the inclusion | at enrollment
  The "Montreal Cognitive Assessment" (MoCA, [23]). The MoCA assesses mild cognitive dysfunctions. It assesses the following functions: short-term memory, visual spatial skills, executive functions, attention, concentration, working memory, language, abstraction skills, calculation and orientation in the time and space. Cognitive impairment is assessed in terms of the score on 30 points (27-30: no cognitive impairment; 18-26: mild; 10-17: moderate; <10: severe). The duration of the test is 20 minutes.
Cognitive efficiency evaluated by the "Montreal Cognitive Assessment" (MOCA) at the end of the following period | at the end of the following period ( i.e. 6 months after the inclusion, 1 month after the end of the MBSR program
  The "Montreal Cognitive Assessment" (MoCA, [23]). The MoCA assesses mild cognitive dysfunctions. It assesses the following functions: short-term memory, visual spatial skills, executive functions, attention, concentration, working memory, language, abstraction skills, calculation and orientation in the time and space. Cognitive impairment is assessed in terms of the score on 30 points (27-30: no cognitive impairment; 18-26: mild; 10-17: moderate; <10: severe). The duration of the test is 20 minutes.
subjective quality of sleep evaluated by the " Pittsburgh Sleep Quality Index " at the inclusion | at enrollment
  This is a self-questionnaire that assesses the subjective quality of sleep in the past month. It includes 19 questions used to calculate 7 components: subjective quality of sleep, sleep latency, sleep duration, sleep efficiency, sleep disturbance, sleep medication, disturbances in daytime functioning. The overall score is obtained by summing the seven components. It ranges from 0: "no difficulty" to 21: "major difficulties".
subjective quality of sleep evaluated by the " Pittsburgh Sleep Quality Index " at the end of the following period | at enrollment
  This is a self-questionnaire that assesses the subjective quality of sleep in the past month. It includes 19 questions used to calculate 7 components: subjective quality of sleep, sleep latency, sleep duration, sleep efficiency, sleep disturbance, sleep medication, disturbances in daytime functioning. The overall score is obtained by summing the seven components. It ranges from 0: "no difficulty" to 21: "major difficulties".
Attentional functions evaluated by the "Test for Attentional Performance" battery (TAP, Zimmerman & Fimm, 2010) at inclusion | at enrollment
  It is a test evaluating the attentional functions (phasic alert, divided attention, sustained attention, visual scanning, intermodal comparison, displacement of the attentional focus, exploration of the visual field / neglect, flexibility, go / nogo, incompatibility, memory of work, eye motility, alertness).
Attentional functions evaluated by the "Test for Attentional Performance" battery (TAP, Zimmerman & Fimm, 2010) at the end of the following period | at the end of the following period ( i.e. 6 months after the inclusion, 1 month after the end of the MBSR program)
  It is a test evaluating the attentional functions (phasic alert, divided attention, sustained attention, visual scanning, intermodal comparison, displacement of the attentional focus, exploration of the visual field / neglect, flexibility, go / nogo, incompatibility, memory of work, eye motility, alertness). The duration of the test is 60 minutes.
Pain evaluated by the Visual Analog Pain Scale (VAS): at the inclusion | at the inclusion visit
  It is a pain self-assessment scale that allows the patient to self-assess the pain experienced by means of a cursor. A slider allows the patient to self-assess the pain felt by means of a cursor. On the front of the slide, a line or pyramid is drawn on which the patient moves the cursor from the "no pain" end to the "maximum pain imaginable" end. On the back of the slide, the caregiver reads the pain felt by the patient using a scale in millimeters (from 0 to 100 mm). Rating is pain absent: 0, mild pain: 1 to 3, moderate pain: 4 to 6, severe pain: 7 to 9, extremely intense pain: 10.
Pain evaluated by the Visual Analog Pain Scale (VAS): at the end of the following period | at the end of the following period ( i.e. 6 months after the inclusion, 1 month after the end of the MBSR program
  It is a pain self-assessment scale that allows the patient to self-assess the pain experienced by means of a cursor. A slider allows the patient to self-assess the pain felt by means of a cursor. On the front of the slide, a line or pyramid is drawn on which the patient moves the cursor from the "no pain" end to the "maximum pain imaginable" end. On the back of the slide, the caregiver reads the pain felt by the patient using a scale in millimeters (from 0 to 100 mm). Rating is pain absent: 0, mild pain: 1 to 3, moderate pain: 4 to 6, severe pain: 7 to 9, extremely intense pain: 10.
Quality of life evaluated by the " Parkinson Disease Quotation " (PDQ-39) at the inclusion | at enrollment
  It is a self-questionnaire in 39 items assessing the quality of life of Parkinson's patients from a motor and psychological point of view, according to the past month. Each question is scored from 0 (no disturbance) to 4 (maximum disturbance). The items are divided into 8 dimensions (activity of daily life, emotional well-being, psychological discomfort, social support, cognitive disorders, communication, physical discomfort, mobility).
Quality of life evaluated by the " Parkinson Disease Quotation " (PDQ-39) at the end of the following period | at the end of the following period ( i.e. 6 months after the inclusion, 1 month after the end of the MBSR program
  It is a self-questionnaire in 39 items assessing the quality of life of Parkinson's patients from a motor and psychological point of view, according to the past month. Each question is scored from 0 (no disturbance) to 4 (maximum disturbance). The items are divided into 8 dimensions (activity of daily life, emotional well-being, psychological discomfort, social support, cognitive disorders, communication, physical discomfort, mobility).
Anxiety evaluated by the " Parkinson Anxiety Scale " (PAS) at the inclusion | at enrollment
  It is a self-questionnaire evaluating anxiety in Parkinson's disease dealing with several dimensions of anxiety: Persistent anxiety (5 items), Episodic anxiety (4 items), Avoidance behavior (3 items) . Each item is rated from 0 (not at all) to 4 (strongly or almost always). The filling time is 5 minutes.
Anxiety evaluated by the " Parkinson Anxiety Scale " (PAS) at the end of the following period | at the end of the following period ( i.e. 6 months after the inclusion, 1 month after the end of the MBSR program
  It is a self-questionnaire evaluating anxiety in Parkinson's disease dealing with several dimensions of anxiety: Persistent anxiety (5 items), Episodic anxiety (4 items), Avoidance behavior (3 items) . Each item is rated from 0 (not at all) to 4 (strongly or almost always). The filling time is 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: François TISON, M.D PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- François TISON, M.D PhD, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No